CLINICAL TRIAL: NCT02920008
Title: A Phase 3, Multicenter, Randomized, Open-Label Study of Guadecitabine (SGI-110) Versus Treatment Choice in Adults With Previously Treated Acute Myeloid Leukemia
Brief Title: Phase 3 Randomized, Open-Label Study of Guadecitabine vs Treatment Choice in Previously Treated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGI-110-06
Record Dates: First submitted 2016-09-28; First posted 2016-09-30 (Estimated); Results first posted 2023-05-25 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML, acute myeloid leukemia, guadecitabine, SGI-110, Phase 3
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- guadecitabine (Experimental): Guadecitabine will be given SC at a dose of 60 mg/m^2 in 28-day cycles (delayed as necessary to allow blood count recovery).
  Interventions: Drug: guadecitabine
- Treatment Choice (TC) (Active Comparator): 1. High intensity
  2. Low intensity
  3. Best supportive care (BSC).
  Interventions: Drug: Treatment Choice (TC)

INTERVENTIONS:
Drug: guadecitabine — In Cycle 1, guadecitabine will be given for 10 days on Days 1-5 and Days 8-12. In Cycle 2, the guadecitabine dose will be 60 mg/m^2 for either 10 days (Days 1-5 and 8-12) or 5 days (Days 1-5 only) based on assessment of disease response, and hematological recovery by Day ≥28.
  Other Names: SGI-110
  Arms: guadecitabine
Drug: Treatment Choice (TC) — * High intensity: intermediate or high dose cytarabine (HiDAC); mitoxantrone, etoposide, and cytarabine (MEC); or fludarabine, cytarabine, G-CSF, +/- idarubicin (FLAG/FLAG-Ida).
  * Low intensity: low dose cytarabine (LDAC), decitabine, or azacitidine.
  * Best Supportive Care (BSC).
  Arms: Treatment Choice (TC)

SUMMARY:
Multicenter, randomized, open-label, parallel-group study of guadecitabine vs treatment choice (TC). Participants will be randomly assigned in a 1:1 ratio to either guadecitabine or TC. TC options include the 8 high or low intensity, locally available regimens below; or Best supportive Care (BSC) alone:

* High intensity (intermediate or high dose cytarabine [HiDAC]; mitoxantrone, etoposide, and cytarabine [MEC]; or fludarabine, cytarabine, granulocyte colony stimulating factor [G-CSF], +/- idarubicin [FLAG/FLAG-Ida]).
* Low intensity (low dose cytarabine [LDAC], decitabine, or azacitidine).
* BSC.

DETAILED DESCRIPTION:
This Phase 3, randomized, open-label, parallel-group multicenter study of the efficacy and safety of guadecitabine in adults with previously treated acute myeloid leukemia (AML) will be conducted in approximately 20 countries. There will be a 14-day screening period, a treatment period, a safety follow-up visit, and a long-term follow-up period. The study is expected to last approximately 2 years. Duration of individual participant participation will vary, and participants may continue to receive treatment for as long as they continue to benefit.

Approximately 404 participants from approximately 100 study centers will be randomly assigned to either guadecitabine or treatment choice (TC) in a 1:1 ratio (approximately 202 participants per group). TC is as follows:

* High intensity: intermediate or high dose cytarabine (HiDAC); mitoxantrone, etoposide, and cytarabine (MEC); or fludarabine, cytarabine, G-CSF, +/- idarubicin (FLAG/FLAG-Ida).
* Low intensity: low dose cytarabine (LDAC), decitabine, or azacitidine.
* Best Supportive Care (BSC).

Guadecitabine will be given subcutaneous (SC) at a dose of 60 microgram per meter square (mg/m^2) in 28-day cycles. In Cycle 1, guadecitabine will be given for 10 days on Days 1-5 and Days 8-12. Cycle 2 will be either the 5-day regimen (Days 1-5) or 10-day regimen (Days 1-5 and 8-12) based on assessment of disease response and hematologic recovery at the end of Cycle 1. In subsequent cycles, guadecitabine treatment will be for 5 days only (Days 1-5).

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants ≥18 years of age who are able to understand study procedures, comply with them, and provide written informed consent before any study-specific procedure.
2. History of cytologically or histologically confirmed diagnosis of AML (except acute promyelocytic leukemia) according to the 2008 World Health Organization (WHO) classification (bone marrow [BM] or peripheral blood [PB] blast counts ≥20%).
3. Performance status (Eastern Cooperative Oncology Group; ECOG) of 0-2.
4. Participants with AML previously treated with initial induction therapy using a standard intensive chemotherapy regimen, including cytarabine and an anthracycline, and who are refractory to initial induction (primary refractory) or in relapse after such initial induction with or without prior HCT.
5. Participants must have either PB or BM blasts ≥5% at time of randomization.
6. Creatinine clearance or glomerular filtration rate ≥30 mL/min as estimated by the Cockroft-Gault (C-G) or other medically acceptable formulas, such as MDRD (Modification of Diet in Renal Disease) or CKD-EPI (the Chronic Kidney Disease Epidemiology Collaboration).
7. Women of child-bearing potential must not be pregnant or breastfeeding and must have a negative pregnancy test at screening. Women of child-bearing potential and men with female partners of child-bearing potential must agree to practice 2 highly effective contraceptive measures of birth control and must agree not to become pregnant or father a child (a) while receiving treatment of guadecitabine, decitabine, or azacitidine and for at least 3 months after completing treatment and (b) while receiving treatment with high-intensity TC or LDAC and for at least 6 months after completing treatment.

Exclusion Criteria:

1. Known clinically active central nervous system (CNS) or extramedullary AML, except leukemia cutis.
2. Participants who are in first relapse after initial induction, if they had a response duration of >12 months from date when first response first documented or if they are good candidates for HCT.
3. BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
4. Second malignancy currently requiring active therapy, except breast or prostate cancer stable on or responding to endocrine therapy.
5. Grade 3 or higher Graft Versus Host Disease (GVHD), or GVHD on either a calcineurin inhibitor or prednisone more than 5 mg/day.
6. Prior treatment with guadecitabine for any indication, or more than 2 cycles of prior decitabine or azacitidine.
7. Hypersensitivity to decitabine, guadecitabine, or any of their excipients.
8. Treated with any investigational therapy within 2 weeks of the first dose of study treatment.
9. Total serum bilirubin >2.5 × upper limit of normal (ULN; except for participants with Gilbert's Syndrome for whom direct bilirubin is <2.5 × ULN), or liver cirrhosis, or chronic liver disease Child-Pugh Class B or C.
10. Known active human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection. Inactive hepatitis carrier status or low viral hepatitis titer on antivirals is allowed.
11. Known significant mental illness or other condition such as active alcohol or other substance abuse or addiction that, in the opinion of the investigator, predisposes the participant to high risk of noncompliance with the protocol.
12. Refractory congestive heart failure unresponsive to medical treatment; active infection resistant to all antibiotics; or non-AML-associated pulmonary disease requiring >2 liters per minute (LPM) oxygen, or any other condition that puts the participant at an imminent risk of death.
13. Participants with high PB blasts >50% AND poor ECOG PS of 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harold N Keer, MD, PhD, Study Director — Astex Pharmaceuticals, Inc.
Locations (95):
- United States (15):
  - University of Southern California, Los Angeles, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - Franciscan Research Center, Indianapolis, Indiana
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medical College, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - University of Oklahoma Medical Center, Oklahoma City, Oklahoma
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - West Virginia University Hospitals, Inc., Morgantown, West Virginia
- Belgium (3):
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Hopital Maisonneuve Rosemont, Montreal
- Denmark (2):
  - Aarhus University Hospital, Aarhus C
  - Rigshospitalet, Copenhagen
- France (9):
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Hôpital de la Conception, Marseille
  - CHRU Montpellier - Saint Eloi, Montpellier
  - Groupe Hospitalier de la Région de Mulhouse et Sud Alsace, Mulhouse
  - Hôpital Saint-Louis, Paris
  - CHU Hopitaux de Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
- Germany (8):
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Marien Hospital Düsseldorf GmbH, Düsseldorf
  - Universitätsklinikum Halle (Saale), Halle
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Medizinischen Fakultät Mannheim der Universität Heidelberg, Mannheim
  - Klinikum der Universität München, München
  - Universitätsklinikum Ulm, Ulm
- Hungary (5):
  - SE ÁOK I. sz. Belgyógyászati Klinika, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Pecsi Tudomanyegyetem Klinikai Központ, Pécs
  - Szegedi Tudományegyetem, Szeged
- Italy (5):
  - IRCCS AOU San Martino - IST, Genova
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele - Milano, Milan
  - A.O.R.N. "A. Cardarelli", Napoli
  - A.S.U Integrata di Udine - Presidio Ospedaliero Santa Maria della Misericordia, Udine
- Japan (17):
  - Akita University Hospital, Akita
  - Chugoku Central Hospital, Fukuyama-Shi
  - Tokai University Hospital, Isehara-shi
  - Saitama Medical Center, Kawagoe-Shi
  - Kobe City Medical Center General Hospital, Kobe
  - Japanese Red Cross Kyoto Daini Hospital, Kyoto
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Gunmaken Saiseikai Maebashi Hospital, Maebashi
  - Nagasaki University Hospital, Nagasaki
  - The Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Kindai University Hospital, Osakasayama-Shi
  - Saga University Hospital, Saga
  - NTT Medical Center Tokyo, Shinagawa-Ku
  - Shizuoka Cancer Center, Shizuoka
  - National Hospital Organization Disaster Medical Center, Tachikawa-Shi
  - Yamagata University Hospital, Yamagata
  - University of Fukui Hospital, Yoshida-Gun
- Instytut Hematologii i Transfuzjologi, Warsaw, Poland
- South Korea (7):
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital (UUH), Ulsan
- Spain (11):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Vall d'Hebron Institut d'Oncologia, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia
- Sahlgrenska University Hospital, Gothenburg, Sweden
- Ukraine (2):
  - Khmelnytskyi Regional Hospital, Khmelnytskyi
  - Poltava Regional Clinical Hospital named after M. V. Sklifosovskoho, Poltava
- United Kingdom (4):
  - Heart of England NHS Foundation Trust - Heartlands Hospital, Birmingham
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology and Oncology Centre, Bristol
  - East Kent Hospitals University NHS Foundation Trust - Kent and Canterbury Hospital, Canterbury
  - St. James's University Hospital, Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roboz GJ, Sanz G, Griffiths EA, Yee K, Kantarjian H, Recher C, Byrne MT, Patkowska E, Kim HJ, Thomas X, Moors I, Stock W, Illes A, Fenaux P, Miyazaki Y, Yamauchi T, O'Connell CL, Hao Y, Keer HN, Azab M, Dohner H. Guadecitabine vs TC in relapsed/refractory AML after intensive chemotherapy: a randomized phase 3 ASTRAL-2 trial. Blood Adv. 2024 Apr 23;8(8):2020-2029. doi: 10.1182/bloodadvances.2023012062. PMID 38231126

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 358 participants were assessed for study inclusion. Of these 56 failed screening assessments. A total of 302 participants were randomized (148 guadecitabine, 154 treatment choice [TC]). Of the randomized participants, 10 did not receive study drug (3 guadecitabine, 7 TC).
Groups:
- Guadecitabine: Guadecitabine was administered subcutaneously (SC) at a dose of 60 milligrams per meter square (mg/m^2) for 10 days on Days 1-5 and Days 8-12 or on Days 1-10 in the first cycle. Second cycle was 60 mg/m^2 for either 10 days (Days 1-5 and 8-12 or Days 1-10) or 5 days (Days 1-5 only) based on assessment of disease response, and hematological recovery by end of Cycle 1. For Cycles ≥3, guadecitabine, 60 mg/m^2 was given for 5 days only (Days 1-5). Each cycle = 28 days.
- Treatment Choice (TC): Intermediate or high dose cytarabine (HiDAC), mitoxantrone, etoposide and cytarabine (MEC) and granulocyte colony-stimulating factors (G-CSF)/fludarabine, cytarabine, G-CSF and idarubicin (FLAG/FLAG-Ida), low dose cytarabine (LDAC), decitabine, azacitidine, or best supportive care (BSC) was administered only. High intensity: Intermediate or HiDAC, recommended as 1-1.5 grams per meter square (g/m^2) every 12 hours or up to 6 g/m^2/day for ≤6 days, maximum 36 g/m^2 per cycle; MEC: For example: mitoxantrone 6-12 mg/m^2 IV (recommended 8 mg/m^2), etoposide 80-200 mg/m^2 intravenous (IV) (recommended 100 mg/m^2), and cytarabine 1000 mg/m^2 IV; each daily for 5 days (Days 1-5); FLAG/FLAG-Ida: For example: fludarabine 25-30 mg/m^2 IV daily Days 1-5; cytarabine 1-2 g/m^2 IV daily for up to 5 days (recommended to be given for 4 hours after fludarabine); G-CSF SC daily from Day 6 up to white cell count recovery with or without idarubicin 8 mg/m^2 IV daily on Days 3 to 5. Low intensity: LDAC 20 mg SC or IV twice daily on Days 1-10; Decitabine 20 mg/m^2 IV daily on Days 1-5; Azacitidine 75 mg/m^2 IV or SC daily on Days 1-7. Best supportive care only.
Period: Overall Study
Arm/Group | Guadecitabine | Treatment Choice (TC)
Started | 148 (Started = Participants who were randomized) | 154
Safety Analysis Set (Safety analysis set included data from all participants randomly assigned to study treatment who received any amount of study treatment or any component of a multi-dose study treatment regimen.) | 145 | 147
Completed | 28 | 20
Not Completed | 120 | 134
Not completed — Death | 117 | 127
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Guadecitabine: Guadecitabine was administered SC at a dose of 60 mg/m^2 for 10 days on Days 1-5 and Days 8-12 or on Days 1-10 in the first cycle. Second cycle was 60 mg/m^2 for either 10 days (Days 1-5 and 8-12 or Days 1-10) or 5 days (Days 1-5 only) based on assessment of disease response, and hematological recovery by end of Cycle 1. For Cycles ≥3, guadecitabine, 60 mg/m^2 was given for 5 days only (Days 1-5). Each cycle = 28 days.
- Treatment Choice (TC): Intermediate or HiDAC, MEC, and FLAG/FLAG-Ida, LDAC, decitabine, azacitidine, or BSC was administered only. High intensity: Intermediate or HiDAC, recommended as 1-1.5 g/m^2 every 12 hours or up to 6 g/m^2/day for ≤6 days, maximum 36 g/m^2 per cycle; MEC: For example: mitoxantrone 6-12 mg/m^2 IV (recommended 8 mg/m^2), etoposide 80-200 mg/m^2 IV (recommended 100 mg/m^2), and cytarabine 1000 mg/m^2 IV; each daily for 5 days (Days 1-5); FLAG/FLAG-Ida: For example: fludarabine 25-30 mg/m^2 IV daily Days 1-5; cytarabine 1-2 g/m^2 IV daily for up to 5 days (recommended to be given for 4 hours after fludarabine); G-CSF SC daily from Day 6 up to white cell count recovery with or without idarubicin 8 mg/m^2 IV daily on Days 3 to 5. Low intensity: LDAC 20 mg SC or IV twice daily on Days 1-10; Decitabine 20 mg/m^2 IV daily on Days 1-5; Azacitidine 75 mg/m^2 IV or SC daily on Days 1-7. Best supportive care only.
- Total: Total of all reporting groups
Arm/Group | Guadecitabine | Treatment Choice (TC) | Total
Number analyzed (Participants) | 148 | 154 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (12.2) | 59.8 (13.1) | 60.8 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 76 | 138
  Male | 86 | 78 | 164
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 16 | 34
  Not Hispanic or Latino | 113 | 114 | 227
  Unknown or Not Reported | 17 | 24 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 95 | 90 | 185
  Black or African American | 3 | 6 | 9
  Asian | 30 | 34 | 64
  American Indian or Alaska Native | 1 | 0 | 1
  Not Reported | 19 | 24 | 43

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival is defined as number of days from day of randomization to date of death, regardless of cause.
Time Frame: From the date of randomization until the date of death, or approximately 34 months
Population: The efficacy analysis set included data from all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 148 | 154
days | 191.0 [141.0 to 253.0] | 163.0 [131.0 to 213.0]
Statistical Analysis 1: Comparison: Guadecitabine vs Treatment Choice (TC); Test type: Superiority; p = 0.3287, Stratified log-rank

2. Secondary Outcome: Event-Free Survival
Description: Event-free survival is defined as number of days from randomization to earliest date of treatment discontinuation (for reasons other than initiation of hematopoietic cell transplant [HCT]), start of alternative anti-leukemia therapy (except HCT), or death.
Time Frame: From the date of randomization until the date of death, or approximately 38 months
Population: The efficacy analysis set included data from all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 148 | 154
days | 90.0 [73.0 to 105.0] | 71.5 [53.0 to 78.0]

3. Secondary Outcome: Long-Term Survival
Description: Survival rate at 1 year after randomization; participants were also followed to estimate 2-year survival rate.
Time Frame: Up to approximately 38 months
Population: The efficacy analysis set included data from all participants randomly assigned to study treatment.
Measure: Number (95% Confidence Interval); unit: proportion
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 148 | 154
proportion
  12-month survival rate | 0.32 [0.25 to 0.40] | 0.26 [0.20 to 0.34]
  24-month survival rate | 0.19 [0.12 to 0.26] | 0.10 [0.05 to 0.17]

4. Secondary Outcome: Number of Days Alive and Out of the Hospital (NDAOH)
Description: Number of days participants alive and out of hospital during first 6 months of the study.
Time Frame: 6 months
Population: The efficacy analysis set included data from all participants randomly assigned to study treatment.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 148 | 154
days | 73.2 [53.2 to 93.2] | 73.9 [53.8 to 94.1]

5. Secondary Outcome: Transfusion Independence Rate
Description: Number of participants without red blood cells (RBC) or platelet transfusion for any 8-week period after treatment divided by total number of participants in efficacy analysis.
Time Frame: Baseline up to approximately 38 months
Population: The efficacy analysis set included data from all participants randomly assigned to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 148 | 154
percentage of participants
  Overall transfusion independence | 20.3 | 13.0
  Platelet transfusion independence | 23.6 | 21.4
  RBC transfusion independence | 21.6 | 14.3

6. Secondary Outcome: Complete Response Rate
Description: The Complete response (CR) rate based on modified International Working Group (IWG) 2003 AML Response Criteria was calculated as the number of participants with a best response of CR divided by the total number of participants included in the efficacy analysis. CR as per modified 2003 IWG AML Response Criteria is absolute neutrophil count (ANC) ≥1000/μL, platelets ≥100,000/μL, independence from red blood cells (RBC) and platelet transfusions over the past week, no leukemic blasts in peripheral blood and bone marrow should contain less than 5% blast cells.
Time Frame: Baseline to end of treatment, or approximately 38 months
Population: The efficacy analysis set included data from all participants randomly assigned to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 148 | 154
percentage of participants | 12.8 | 7.1

7. Secondary Outcome: Combined Complete Response and Complete Response With Partial Hematologic Recovery Rate
Description: The combined CR and CR with partial hematologic recovery rate based on modified International Working Group (IWG) 2003 AML Response Criteria was calculated as number of participants with CR and CR with partial hematologic recovery divided by the total number of participants included in the efficacy analysis. CR as per modified 2003 IWG AML Response Criteria is absolute neutrophil count (ANC) ≥1000/μL, platelets ≥100,000/μL, independence from red blood cells (RBC) and platelet transfusions over the past week, no leukemic blasts in peripheral blood and bone marrow should contain less than 5% blast cells.
Time Frame: Baseline to end of treatment, or approximately 38 months
Population: The efficacy analysis set included data from all participants randomly assigned to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 148 | 154
percentage of participants | 16.9 | 7.8

8. Secondary Outcome: Composite Complete Response Rate
Description: Composite complete response rate based on modified IWG 2003 AML Response Criteria defined as number of participants with best response of CR, CR with incomplete platelet recovery (CRp), or CR with incomplete blood count recovery (CRi) divided by total number of participants in efficacy analysis. CR as per modified 2003 IWG AML Response Criteria is ANC ≥1000/μL, platelets ≥100,000/μL, independence from RBC and platelet transfusions over the past week, no leukemic blasts in peripheral blood and bone marrow should contain less than 5% blast cells. CRp is defined as ANC ≥1000/μL, Platelets <100,000/μL, independence from RBC transfusions over the past week, no leukemic blasts and bone marrow should contain less than 5% blast cells. CRi is defined as ANC <1000/μL, no leukemic blasts and bone marrow should contain less than 5% blast cells.
Time Frame: Baseline to end of treatment, or approximately 38 months
Population: The efficacy analysis set included data from all participants randomly assigned to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 148 | 154
percentage of participants | 27.0 | 14.3

9. Secondary Outcome: Hematopoietic Cell Transplant (HCT) Rate
Description: Number of participants who received HCT after randomization divided by total number of participants in efficacy analysis.
Time Frame: Baseline to long term follow-up or approximately 38 months
Population: The efficacy analysis set included data from all participants randomly assigned to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 148 | 154
percentage of participants | 17.6 | 16.2

10. Secondary Outcome: Duration of Complete Response (CR) + CR With Partial Hematologic Recovery (CRh)
Description: The time from first CR or CRh to time of relapse (the date of the earliest of the following 3 events):
  1. relapse (defined as the earliest time point whereby BM assessment or PB assessment by the investigator indicate relapse/disease progression due to confirmed reappearance of leukemic blasts in PB or ≥5% leukemic blasts in BM, or clinical progression determined by the investigator),
  2. start of alternative therapy (except HCT) or
  3. death.
Time Frame: Baseline to end of treatment, or approximately 38 months
Population: The efficacy analysis set included data from all participants randomly assigned to study treatment.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 25 | 12
days | 124 [73.0 to 315.0] | 63 [8.0 to 71.0]

11. Secondary Outcome: Change From Baseline in EuroQoL-5 Dimension 5 Level (EQ-5D-5L) Index Scores
Description: Index score is calculated based on 5-level version of the EQ-5D descriptive system using the value set for England.
  The range of index score is from -0.281 (for the worst health state, score of 5 for all categories) to 1 (for the best health state, score of 1 for all categories).
Time Frame: Baseline to 6 months
Population: The efficacy analysis set included data from all participants randomly assigned to study treatment. Overall number of participants analyzed is the number of participants with data available for analysis in this outcome measure.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 107 | 102
score on a scale
  Cycle 2 Day 1 | -0.027 [-0.061 to 0.007] | -0.034 [-0.068 to 0.001]
  Cycle 3 Day 1: number analyzed (Participants) | 80 | 77
  Cycle 3 Day 1 | -0.026 [-0.063 to 0.011] | -0.028 [-0.066 to 0.010]
  Cycle 4 Day 1: number analyzed (Participants) | 71 | 55
  Cycle 4 Day 1 | -0.008 [-0.050 to 0.034] | -0.061 [-0.108 to -0.015]
  Cycle 5 Day 1: number analyzed (Participants) | 57 | 48
  Cycle 5 Day 1 | -0.022 [-0.072 to 0.027] | -0.072 [-0.126 to -0.019]
  Cycle 6 Day 1: number analyzed (Participants) | 48 | 38
  Cycle 6 Day 1 | -0.027 [-0.071 to 0.017] | -0.070 [-0.188 to -0.022]
  Cycle 7 Day 1: number analyzed (Participants) | 37 | 31
  Cycle 7 Day 1 | -0.020 [-0.071 to 0.030] | -0.022 [-0.076 to 0.033]

12. Secondary Outcome: Change in EQ-5D-5L Visual Analogue Scale (VAS) Score
Description: VAS score is obtained using vertical 20-cm visual analogue scale with the top value of 100 labelled as 'the best health you can imagine' and the bottom value of 0 labelled as 'the worst health you can imagine'.
Time Frame: Baseline to 6 months
Population: as for outcome 11
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 107 | 102
score on a scale
  Cycle 2 Day 1 | -2.80 [-6.26 to 0.65] | -1.86 [-5.40 to 1.67]
  Cycle 3 Day 1: number analyzed (Participants) | 80 | 77
  Cycle 3 Day 1 | -0.61 [-4.08 to 2.87] | -1.47 [-5.02 to 2.08]
  Cycle 4 Day 1: number analyzed (Participants) | 71 | 56
  Cycle 4 Day 1 | 1.13 [-2.24 to 4.51] | -2.37 [-6.04 to 1.29]
  Cycle 5 Day 1: number analyzed (Participants) | 57 | 48
  Cycle 5 Day 1 | 1.28 [-2.88 to 5.44] | -2.30 [-6.83 to 2.22]
  Cycle 6 Day 1: number analyzed (Participants) | 47 | 38
  Cycle 6 Day 1 | 0.67 [-3.51 to 4.85] | -1.42 [-6.04 to 3.21]
  Cycle 7 Day 1: number analyzed (Participants) | 37 | 31
  Cycle 7 Day 1 | -0.44 [-5.66 to 4.78] | -0.77 [-6.46 to 4.93]

13. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can therefore be any unfavorable and unintended sign (including a clinically significant abnormal finding in laboratory tests or other diagnostic procedures), symptom, or disease temporally associated with the use of a drug, without any judgment about causality.
Time Frame: From first dose until 30 days after the last dose of study drug, or approximately 38 months
Population: The safety analysis set included data from all participants randomly assigned to study treatment who received any amount of study treatment or any component of a multi-dose study treatment regimen.
Measure: Number; unit: percentage of participants
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 145 | 147
percentage of participants | 96.6 | 97.3

14. Secondary Outcome: All-Cause Mortality
Description: All-cause mortality in the first 30 days and first 60 days after the start of treatment divided by the total number of participants receiving at least one dose of study treatment.
Time Frame: From the first dose until 60 days after the first dose of study drug
Population: The efficacy analysis set included data from all participants randomly assigned to study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Guadecitabine | Treatment Choice (TC)
Number analyzed (Participants) | 145 | 147
percentage of participants
  Within 30 days: number analyzed (Participants) | 17 | 14
  Within 30 days | 11.7 | 9.5
  Within 60 days: number analyzed (Participants) | 36 | 30
  Within 60 days | 24.8 | 20.4

ADVERSE EVENTS:
Time Frame: From first dose until 30 days after the last dose of study drug, or approximately 38 months
Description: All-cause mortality is reported for enrolled participants in the study. The serious and other adverse events is reported for safety analysis set which included data from all participants randomly assigned to study treatment who received any amount of study treatment or any component of a multi-dose study treatment regimen.
Arm/Group | Guadecitabine | Treatment Choice (TC)
All-Cause Mortality (participants affected / at risk) | 117/148 | 129/154
Serious Adverse Events (participants affected / at risk) | 113/145 | 91/147
Other Adverse Events (participants affected / at risk) | 138/145 | 137/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guadecitabine (N=145) | Treatment Choice (TC) (N=147)
Embolism (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Asthenia (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 2 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 6
Suicidal ideation (Psychiatric disorders) | 1 | 0
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 1
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Troponin T increased (Investigations) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 4 | 0
Cardiac failure (Cardiac disorders) | 3 | 1
Cardiac failure acute (Cardiac disorders) | 2 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 2
Aplasia (Congenital, familial and genetic disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 4 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 41 | 33
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2
Brain stem infarction (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 2 | 2
Hydrocephalus (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Oesophageal mucosal tear (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 1
Tongue oedema (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 2 | 2
Anal infection (Infections and infestations) | 1 | 1
Anorectal infection (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 4 | 5
Bartholinitis (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 4 | 0
Cellulitis (Infections and infestations) | 4 | 2
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Corynebacterium bacteraemia (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Dermo-hypodermitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 4 | 3
Disseminated varicella zoster vaccine virus infection (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Ecthyma (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0
Enterobacter infection (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
External ear cellulitis (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Genital infection (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Infective myositis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Intestinal sepsis (Infections and infestations) | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 1 | 1
Liver abscess (Infections and infestations) | 1 | 0
Mucormycosis (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Parvovirus B19 infection (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 27 | 25
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 15 | 16
Septic shock (Infections and infestations) | 7 | 5
Sinusitis fungal (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 3
Staphylococcal bacteraemia (Infections and infestations) | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 2 | 2
Streptococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Guadecitabine (N=145) | Treatment Choice (TC) (N=147)
Hypertension (Vascular disorders) | 15 | 4
Hypotension (Vascular disorders) | 19 | 11
Asthenia (General disorders) | 11 | 15
Fatigue (General disorders) | 20 | 27
Injection site reaction (General disorders) | 29 | 12
Oedema peripheral (General disorders) | 23 | 23
Pyrexia (General disorders) | 33 | 36
Insomnia (Psychiatric disorders) | 14 | 13
Contusion (Injury, poisoning and procedural complications) | 11 | 6
Alanine aminotransferase increased (Investigations) | 12 | 7
Aspartate aminotransferase increased (Investigations) | 11 | 8
Blood alkaline phosphatase increased (Investigations) | 6 | 8
Blood bilirubin increased (Investigations) | 8 | 9
Blood creatinine increased (Investigations) | 8 | 4
Weight decreased (Investigations) | 5 | 9
Anaemia (Blood and lymphatic system disorders) | 37 | 41
Febrile neutropenia (Blood and lymphatic system disorders) | 25 | 29
Leukopenia (Blood and lymphatic system disorders) | 14 | 14
Neutropenia (Blood and lymphatic system disorders) | 47 | 28
Thrombocytopenia (Blood and lymphatic system disorders) | 43 | 46
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 9
Dizziness (Nervous system disorders) | 8 | 11
Headache (Nervous system disorders) | 30 | 20
Abdominal pain (Gastrointestinal disorders) | 11 | 11
Constipation (Gastrointestinal disorders) | 33 | 33
Diarrhoea (Gastrointestinal disorders) | 36 | 32
Dyspepsia (Gastrointestinal disorders) | 12 | 5
Haemorrhoids (Gastrointestinal disorders) | 11 | 9
Nausea (Gastrointestinal disorders) | 42 | 38
Stomatitis (Gastrointestinal disorders) | 16 | 20
Vomiting (Gastrointestinal disorders) | 24 | 20
Dysuria (Renal and urinary disorders) | 8 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 12 | 7
Rash (Skin and subcutaneous tissue disorders) | 11 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 7
Decreased appetite (Metabolism and nutrition disorders) | 27 | 20
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 29 | 38
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 | 16
Hyponatraemia (Metabolism and nutrition disorders) | 10 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 13 | 9
Oral herpes (Infections and infestations) | 8 | 5
Pneumonia (Infections and infestations) | 15 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/08/NCT02920008/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT02920008/SAP_001.pdf